CLINICAL TRIAL: NCT06360094
Title: A Phase IIa/IIb, Randomised, Double Blind, Placebo-controlled, Parallel-group Dose-finding Study to Examine the Efficacy and Safety of BI 1839100 Administered Orally Over a 12-week Treatment Period in Patients With Idiopathic Pulmonary Fibrosis or Progressive Pulmonary Fibrosis With Clinically Meaningful Cough
Brief Title: A Study to Test Whether BI 1839100 Improves Cough in People With Idiopathic Pulmonary Fibrosis or Progressive Pulmonary Fibrosis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1490-0004; 2023-510249-79-00 (Registry Identifier: CTIS); U1111-1301-1311 (Registry Identifier: WHO Registry (ICTRP))
Record Dates: First submitted 2024-04-08; First posted 2024-04-11 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Idiopathic Pulmonary Fibrosis; Progressive Pulmonary Fibrosis
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Phase IIa/IIb, IPF cohort: Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Phase IIa/IIb, IPF cohort: BI 1839100 low dose (Experimental)
  Interventions: Drug: BI 1839100
- Phase IIa/IIb, IPF cohort: BI 1839100 medium dose (Experimental)
  Interventions: Drug: BI 1839100
- Phase IIa/IIb, IPF cohort: BI 1839100 high dose (Experimental)
  Interventions: Drug: BI 1839100
- Phase IIb, PPF cohort: Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Phase IIb, PPF cohort: BI 1839100 high dose (Experimental)
  Interventions: Drug: BI 1839100

INTERVENTIONS:
Drug: BI 1839100 — BI 1839100
  Arms: Phase IIa/IIb, IPF cohort: BI 1839100 high dose; Phase IIa/IIb, IPF cohort: BI 1839100 low dose; Phase IIa/IIb, IPF cohort: BI 1839100 medium dose; Phase IIb, PPF cohort: BI 1839100 high dose
Drug: Placebo — Placebo
  Arms: Phase IIa/IIb, IPF cohort: Placebo; Phase IIb, PPF cohort: Placebo

SUMMARY:
Adults 40 years of age and older with idiopathic pulmonary fibrosis (IPF) or 18 years and older with progressive pulmonary fibrosis (PPF) can participate in this study. Only people who have a chronic cough can take part. The purpose of this study is to find out how well BI 1839100 helps reduce coughing in people with IPF or PPF.

Participants who have IPF are put into 4 groups by chance. Participants in 3 groups get different doses of BI 1839100. Participants in 1 group get placebo. Placebo looks like BI 1839100 but does not contain any medicine. Participants take the treatment for 3 months. After 1 month of treatment, participants who take the highest dose will have coughing measured to find out if the medicine works. If it does not work, the study may be stopped. Participants who have IPF are in the study for slightly longer than 4 months. During this time, they visit the study site 7 times. This study will also measure the effects of BI 1839100 on coughing and lung function in a smaller group of people with PPF.

During the study, coughing is measured over 24 hours about once per month using a portable device given to participants to use during the study. Participants fill in questionnaires about their coughing. Doctors also perform breathing tests that measure how well the lungs are working at the site visits. Researchers compare the results between participants who take BI 1839100 and placebo. The doctors also regularly check participants' health and take note of any unwanted effects.

ELIGIBILITY:
Inclusion Criteria

For Idiopathic Pulmonary Fibrosis (IPF) cohort:

* Minimum age: 40 years
* Diagnosis of IPF
* Chronic cough (>8 weeks prior to Visit 1) attributed to IPF and refractory to treatment for known causes (Principal Investigator (PI) assessment)
* Cough Severity visual analogue scale (VAS) ≥30 mm at Visit 1 and Visit 2B
* Forced vital capacity (FVC) ≥45% of predicted normal at Visit 1
* Diffusing capacity of the lungs for carbon monoxide (DLCO) >25% of predicted normal at Visit 1
* Patients may be either:

  * On stable therapy with nintedanib or pirfenidone for ≥12 weeks prior to Visit 1 and are planning to stay on this background treatment for the whole trial duration. Combination of nintedanib plus pirfenidone will not be allowed
  * Not on therapy with nintedanib or pirfenidone for ≥12 weeks prior to Visit 1 (either antifibrotic (AF)-treatment naïve or previously discontinued) and do not plan to start or re-start AF treatment during the trial. It is not permitted to delay nintedanib or pirfenidone therapy for the purpose of participating in this trial
* Patients aged ≥40 years when signing the informed consent

For Progressive Pulmonary Fibrosis (PPF) cohort:

* Minimum age: 18 years
* Diagnosis of PPF
* Chronic cough (>8 weeks prior to Visit 1) attributed to PPF, refractory to treatment for known causes (PI assessment)
* Cough Severity VAS ≥30 mm at Visit 1 and Visit 2B
* FVC ≥45% of predicted normal at Visit 1
* DLCO ≥25% of predicted normal at Visit 1
* If receiving immunomodulatory therapy for interstitial lung disease (ILD), allowed medications include tacrolimus, mycophenolate mofetil, or azathioprine (stable dose for 12 weeks prior to Visit 1)
* Patients may be either:

  * On a stable therapy with nintedanib for ≥12 weeks prior to Visit 1 and are planning to stay on this background treatment for the whole trial duration
  * Not on a therapy with nintedanib for ≥12 weeks prior to Visit 1 (either AF-treatment naïve or previously discontinued) and do not plan to start or re-start AF treatment during the trial. It is not permitted to delay nintedanib or pirfenidone therapy for the purpose of participating in this trial
* Patients aged >18 years when signing the informed consent Further inclusion criteria apply.

Exclusion criteria for IPF and PPF cohorts:

* Acute exacerbation of IPF/PPF within 12 weeks prior to Visit 1
* Forced expiratory volume in 1 second (Forced expiratory volume in 1 second (FEV1))/FVC <0.7 at Visit 1
* Known reversible airflow obstruction/response to bronchodilators
* In the opinion of the Investigator, other clinically significant pulmonary abnormalities, including primary bronchitic and bronchiectatic disorder
* Upper or lower respiratory tract infection within 4 weeks prior to Visit 1
* Ongoing chronic pulmonary infection (e.g. mycobacterial or fungal disease)
* Current smokers (tobacco use within the 6 months prior to Visit 1)
* Initiation or change in supplemental oxygen requirement during 4 weeks prior to Visit 1 Further exclusion criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2024-08-28 (Actual); Primary Completion 2025-09-02 (Actual); Study Completion 2025-09-02 (Actual)

PRIMARY OUTCOMES:
IPF cohort - Phase IIa: Change from baseline in 24-h cough frequency (Cough count (CC)/h) | At baseline, at week 4
IPF cohort - Phase IIb: Change from baseline in 24-h cough frequency (CC/h) | At baseline, at week 12

SECONDARY OUTCOMES:
IPF cohort - Phase IIa: Absolute change from baseline in Cough Severity Numerical rating scale (NRS) score | At baseline, at week 4
  NRS: a single-item patient reported outcome measure to assess cough severity on a 11-point numerical rating scale ranging from 0 (no cough) to 10 (worst possible cough) with a recall period of the past 7 days. Higher scores indicate higher severity of cough.
IPF cohort - Phase IIa: Absolute change from baseline in Cough Severity Visual analogue scale (VAS) score (mm) | At baseline, at week 4
  VAS: the cough severity VAS is scored according to the distance between no cough (0) and the mark set by the participant, with higher distance indicating higher severity of cough.
IPF cohort - Phase IIb: Cough responder status, defined as a ≥30% reduction in 24-h cough frequency (CC/h) | At baseline, at week 12
IPF cohort - Phase IIb: Absolute change from baseline in Forced vital capacity (FVC) (mL) | At baseline, at week 12
IPF cohort - Phase IIb: Absolute change from baseline in Cough Severity NRS score | At baseline, at week 12
IPF cohort - Phase IIb: Absolute change from baseline in Cough Severity VAS score (mm) | At baseline, at week 12
IPF cohort - Phase IIb: Absolute change from baseline in Living with Pulmonary Fibrosis (L-PF) symptom cough domain score | At baseline, at week 12
  L-PF: the L-PF symptom module domain and total scores as well as the L-PF impact module total score ranges from 0 to 100, with higher scores indicating a greater impairment.
IPF cohort - Phase IIb: Absolute change from baseline in Leicester Cough Questionnaire (LCQ) physical domain score | At baseline, at week 12
  LCQ: the total score ranges from 3 to 21. A higher score indicates better cough specific quality of life.

CONTACTS AND LOCATIONS:
Locations (99):
- United States (18):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Critical Care, Pulmonary and Sleep Associates, Lakewood, Colorado
  - Clinical Research Specialists LLC - Kissimmee, Kissimmee, Florida
  - The Iowa Clinic, PC, West Des Moines, Iowa
  - Advanced Pulmonary Research, Warren, Michigan
  - Memorial Hospital Gulfport, Gulfport, Mississippi
  - Northern Westchester Hospital, Mount Kisco, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Columbia University Medical Center-New York Presbyterian Hospital, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Coastal Carolina Health Care, P.A. Pulmonary and Sleep Medicine, New Bern, North Carolina
  - Southeastern Research Center-Winston Salem-69289, Winston-Salem, North Carolina
  - Clinical Research Associates of Central PA, DuBois, Pennsylvania
  - Temple University Hospital, Philadelphia, Pennsylvania
  - Lowcountry Lung and Critical Care, Charleston, South Carolina
  - Spartanburg Medical Research, Spartanburg, South Carolina
  - A & A Research Consultants, LLC, Edinburg, Texas
  - Pulmonary Associates of Richmond, Inc., Richmond, Virginia
- Australia (2):
  - Launceston Respiratory & Sleep Centre, Launceston, Tasmania
  - Lung Research Victoria, Footscray, Victoria
- CHR de la Citadelle, Liège, Belgium
- Canada (3):
  - Gordon & Leslie Diamond Health Care Centre (UBC), Vancouver, British Columbia
  - St. Joseph's Healthcare Hamilton, Hamilton, Ontario
  - Centre Hospitalier de l'Universite de Montreal (CHUM), Montreal, Quebec
- China (11):
  - The Second Xiangya Hospital Of Central South University, Changsha
  - West China Hospital of Sichuan University, Chengdu
  - People's Hospital of Sichuan Province, Chengdu
  - First Affiliated Hospital of Guangzhou Medical University, Guangzhou
  - Zhejiang Hospital, Hangzhou
  - Anhui Provincial Hospital, Hefei
  - Nanjing Drum Tower Hospital, Nanjing
  - Shanghai Pulmonary Hospital, Shanghai
  - China Shenyang Chest Hospital, Shenyang
  - Tianjin Medical University General Hospital, Tianjin
  - Affiliated Hospital, Xuzhou Medical college, Xuzhou
- University Thomayer´s Hospital, Prague, Czechia
- Odense University Hospital, Odense, Denmark
- Finland (3):
  - HYKS Keuhkosairauksien tutkimusyksikkö, Helsinki
  - Oulun yliopistollinen keskussairaala, Oulu
  - TYKS, Turku
- France (6):
  - HOP d'Angers, Angers
  - HOP Avicenne, Bobigny
  - HOP CHU Caen, Caen
  - HOP Michallon, La Tronche
  - HOP Nord Laennec, Nantes
  - HOP Bretonneau, Tours
- Germany (7):
  - Universitätsklinikum Aachen, AöR, Aachen
  - CIMS Studienzentrum Bamberg GmbH, Bamberg
  - Ruhrlandklinik, Westdeutsches Lungenzentrum am Universitätsklinikum Essen gGmbH, Essen
  - Universitätsklinikum Freiburg, Freiburg im Breisgau
  - Medizinische Hochschule Hannover, Hanover
  - Thoraxklinik-Heidelberg gGmbH am Universitätsklinikum Heidelberg, Heidelberg
  - Krankenhaus Bethanien gGmbH, Solingen
- Greece (2):
  - Hospital of Heraklion (PAGNI), Crete
  - Univ. Gen. Hosp. of Patras, Pátrai
- Italy (4):
  - Ospedale Classificato San Giuseppe, Milan
  - Azienda Ospedaliera Universitaria di Padova, Padua
  - Pol. Universitario Tor Vergata, Roma
  - Fondazione Policlinico Universitario A. Gemelli IRCCS, Roma
- Japan (9):
  - University of Fukui Hospital, Fukui, Yoshida-gun
  - National Hospital Organization Kyushu Medical Center, Fukuoka, Fukuoka
  - Kyushu University Hospital, Fukuoka, Fukuoka
  - Sapporo Medical University Hospital, Hokkaido, Sapporo
  - National Hospital Organization Himeji Medical Center, Hyogo, Himeji
  - Kanagawa Cardiovascular and Respiratory Center, Kanagawa, Yokohama
  - Tokushima University Hospital, Tokushima, Tokushima
  - Toho University Omori Medical Center, Tokyo, Ota-ku
  - National Center for Global Health and Medicine, Tokyo, Shinjuku-ku
- Malaysia (2):
  - Hospital Sultan Idris Shah Serdang, Kajang
  - Institut Perubatan Respiratori, Kuala Lumpur
- Netherlands (2):
  - Amphia Ziekenhuis, Breda
  - Erasmus Medisch Centrum-ROTTERDAM-50697, Rotterdam
- New Zealand (3):
  - Christchurch Hospital, Christchurch
  - Waikato Hospital, Hamilton
  - Greenlane Clinical Centre, One Tree Hill, Auckland
- Norway (3):
  - Haukeland Universitetssykehus, Bergen
  - Akershus Universitetssykehus HF, Lørenskog
  - Oslo Universitetssykehus HF, Rikshospitalet, Oslo
- Singapore General Hospital, Singapore, Singapore
- South Korea (2):
  - Inje University Sanggye Paik Hospital, Seoul
  - Asan Medical Center, Seoul
- Spain (5):
  - Hospital Universitari Vall D Hebron, Barcelona
  - Hospital de Galdakao, Galdakao
  - Hospital Universitario Virgen de la Victoria, Málaga
  - Hospital Central de Asturias, Oviedo
  - Hospital Quirónsalud Madrid, Pozuelo de Alarcón
- Sweden (2):
  - Skånes universitetssjukhus, Lund, Lund
  - CTC Clinical Trial Consultants AB, Uppsala
- Taiwan (2):
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - Taichung Veterans General Hospital, Taichung
- Thailand (4):
  - Chulalongkorn Hospital, Bangkok
  - Srinagarind Hospital, Khon Kaen
  - Ramathibodi Hospital, Ratchatewi
  - Songklanagarind Hospital, Songkhla
- United Kingdom (5):
  - Royal Devon and Exeter Hospital, Wonford, Exeter
  - Royal Lancaster Infirmary, Lancaster
  - Royal Brompton Hospital, London
  - Wythenshawe Hospital, Manchester
  - Southampton General Hospital, Southampton

IPD SHARING:
Plan to Share IPD: Yes
Once the criteria in section "Time Frame" are fulfilled, researchers can use the following link https://www.mystudywindow.com/msw/datasharing to request access to the clinical study documents regarding this study, and upon a signed "Document Sharing Agreement".
  Furthermore, researchers can request access to the clinical study data, for this and other listed studies, after the submission of a research proposal and according to the terms outlined in the website.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: One year after the approval has been granted by major Regulatory Authorities and after the primary manuscript has been accepted for publication, or after termination of the development program.
Access Criteria: For study documents - upon signing of a 'Document Sharing Agreement'.
  For study data - 1. after the submission and approval of the research proposal (checks will be performed by the sponsor and/or the independent review panel, including checking that the planned analysis does not compete with sponsor's publication plan); 2. and upon signing of a legal agreement.
URL: https://www.mystudywindow.com/msw/datasharing

REFERENCES:
- See also: Related Info — https://www.mystudywindow.com